CLINICAL TRIAL: NCT02475603
Title: Clinical, Biochemical and Neurophysiological Consequences of Intraoperative
Brief Title: Clinical, Biochemical and Neurophysiological Consequences of Intraoperative Tourniquet During Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Ahmed Jawhar, Dr, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012-334N-MA
Record Dates: First submitted 2015-06-10; First posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2012-09

CONDITIONS: Muscles Ischemia
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tourniquet (Experimental): Total knee arthroplasty will be performed with tourniquet
  Interventions: Procedure: Total knee arthroplasty
- non-tourniquet (Experimental): Total knee arthroplasty will be performed without tourniquet
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Total knee arthroplasty

SUMMARY:
Clinical, Biochemical and Neurophysiological Consequences of Intraoperative Tourniquet During Total Knee Arthroplasty:

WOMAC-Score Knee-Score Radiographic Evaluations and Scoring System Biochemical muscle biopsy analysis

DETAILED DESCRIPTION:
Biochemistry: Analysis of the muscles biopsies Clinical: Bloodloss, Complications, WOMAC-Score, Knee-Score Radiographics: Evaluations and Scoring System Neurophysiology Evaluation of N. femoralis

ELIGIBILITY:
Inclusion Criteria:

* Age = 55-85 years
* Osteoarthritis of knee joint (degree III or IV)
* Physical status (ASA I or II)
* Body mass index < 45 kg/m²
* Written informed consent

Exclusion Criteria:

* Age <55 or > 85years
* Osteoarthritis knee joint (degree I or II)
* Physical status (ASA III or IV)
* Body mass index ≥ 45 kg/m²
* Unable to provide written consent
* Malignant disease
* Rheumatoid disease
* Infectious disease
* Coagulation disorder
* History of deep vein thrombosis or pulmonary embolism
* Peripheral arterial disease
* Immune deficiency
* Medication (Glucocorticoid, Aspirin, Heparin, Cumardine, Wafarin)
* Neurological dysfunction
* Liver insufficiency
* Coronary heart disease
* Immobility

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical Data | During operation 60 min Ischemia/Shame-Ischemia Time
  Measurement of intracellular proteolytic activity

SECONDARY OUTCOMES:
Bloodloss | 1 week postoperative
Complications | 6 months postoperative
Clinical Scores | 6 months postoperative
  WOMAC-Score, Knee-Score
Radiographic Scores | 1 Week postoperative
  Prosthesis Position on radiographs
Electrophysiological Evaluation of the N. femoralis | 1 Week postoperative
  Nerve function analysis

CONTACTS AND LOCATIONS:
Overall Officials: Udo Obertacke, Prof. Dr., Study Director — UMM
Locations (1):
- UMM, Mannheim, Badenwürtemberg, Germany

REFERENCES:
- [Background] Girard N. Evidence appraisal of Zhang W, Li N, Chen S, Tan Y, Al-Aidaros M, Chen L. The effects of a tourniquet used in total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2014;9(1):13. http://www.josr-online.com/content/9/1/13. Accessed May 30, 2014. AORN J. 2014 Aug;100(2):224-8. doi: 10.1016/j.aorn.2014.06.003. No abstract available. PMID 25219028
- [Derived] Jawhar A, Skeirek D, Stetzelberger V, Kollowa K, Obertacke U. No effect of tourniquet in primary total knee arthroplasty on muscle strength, functional outcome, patient satisfaction and health status: a randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2020 Apr;28(4):1045-1054. doi: 10.1007/s00167-019-05646-5. Epub 2019 Aug 1. PMID 31372679